CLINICAL TRIAL: NCT03554720
Title: Radiostereometric Analysis (RSA) of the ATTUNE Knee System: A Randomized Controlled Trial Comparing Traditional Versus Enhanced-Fixation Device Designs
Brief Title: RSA of the ATTUNE Knee System: RCT Comparing Traditional Vs Enhanced-Fixation Device Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Collaborators: Orthopaedic Innovation Centre (Other); Dalhousie University (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS21601
Record Dates: First submitted 2018-05-18; First posted 2018-06-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard implants (Active Comparator): ATTUNE PS Knee
  Interventions: Device: ATTUNE PS Knee
- Enhanced-Fixation (Active Comparator): ATTUNE S+ PS Knee
  Interventions: Device: ATTUNE S+ PS Knee

INTERVENTIONS:
Device: ATTUNE PS Knee — The ATTUNE PS Knee is the standard implants.
  Arms: Standard implants
Device: ATTUNE S+ PS Knee — The ATTUNE S+ PS Knee is the enhanced fixation.
  Arms: Enhanced-Fixation

SUMMARY:
The principal objective of this study is to compare migration patterns between the Attune and Attune S+ PS knee systems using model-based RSA over the first 2 post-operative years. Secondary objectives include; comparison of 2-year migration values against published thresholds for adequate short-term fixation, quantify changes in functional and health status of subjects following surgery and compare between study groups, and assess occurrences of complications following surgery.

DETAILED DESCRIPTION:
This is a multi-centre, randomized controlled trial of patients undergoing posterior-stabilized total knee arthroplasty. In this study, the investigators propose to randomize 50 subjects to receive either the standard Attune PS TKA (n=25) or the enhanced fixation Attune S+ PS TKA (n=25) and follow them for a period of 2 years post-operatively. The primary outcome of the study will be stability of fixation of the tibial baseplate as measured by model-based RSA. Secondary outcomes will be to determine the functionality of patients after surgery using self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating primary total knee arthroplasty
* Between the ages of 21 and 80 inclusive
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection
* Medical condition precluding major surgery

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
RSA Migration | 2 Years
  Migration of the tibial and femoral components between the 2 device designs.

SECONDARY OUTCOMES:
Knee Replacement Expectation Survey (KRES) | Preoperative
  The KRES is a patient reported questionnaire that consists of 19 questions. The questions ask how each expectation is important in the treatment of the knee. The scale is rated: 1 (Very important) to 5 (This does not apply to me). The score ranges from 19 to 95 with higher scores associated with higher expectations.
European Quality of Life (EQ-5D-5L) | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in functional outcomes assessments. The EuroQol 5D 5L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Pain score | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported satisfaction as measured using the visual analogue scale (VAS) from 0 (No pain) - 100 (Worst pain imaginable)
Patient satisfaction | Preoperative, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported pain severity as measured using the visual analogue scale (VAS) from 0 (Unsatisfied) - 100 (Completely satisfied)
Oxford 12 Knee | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in functional outcomes assessments, patient reported outcome
University of California at Los Angeles (UCLA) Activity Level scale | Preoperative, 6 Months, 1 Year and 2 Years]
  Evaluate and compare the change in UCLA activity score compared to baseline in the study cohort. UCLA activity scores range from 1 to 10, and is a measure of activity with 10 being most active.
Pain Catastrophizing Scale (PCS) | Preoperative and 1 Year
  The patient are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain. Each PCS item is rated on a 5-point scale: 0 (not at all) to 4 (all the time). The PCS total score is computed by summing responses to the 13 items. PCS total scores range from 0 - 52.
Pre-operative Patient's Knee Implant Performance (PKIP) | Preoperative, 6 Months, 1 Year and 2 Years
  The Pre-surgical and/or Post-surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient reported questionnaire that consists of 24 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likaert- like response option.
Patient complications | Preoperative, 1 Week, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate the type and frequency of the complications/adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD MPH FRCSC, Principal Investigator — University of Manitoba; Glen Richardson, MD MSc FRCSC, Principal Investigator — Dalhousie University; Douglas Naudie, MD FRCSC, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - Concordia Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario